CLINICAL TRIAL: NCT07035561
Title: Rituximab Therapy in Patients With Treatment Refractory Hypersenstivity Pneumonitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shereen Medhat Mohammed Elsayed Nassar (Other)
Responsible Party: Sponsor-Investigator, Shereen Medhat Mohammed Elsayed Nassar, Shereen Medhat Mohammed Elsayed Nassar was the principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-180-2023; MD-180-2023 (Other: Cairo University Hospitals)
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypersenstivity Pneumonitis; ILD
Keywords: Rituximab; FVC; Hypersenstivity Pneumonitis; treatment
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: * Rituximab will be administered by an intravenous infusion.
  * Two doses of Rituximab will be given, the first dose at day 0 and the second dose at day 15, 1 gram of Rituximab will be given in each dose.
  * Patients will be given acetaminophen and antihistamine before each infusion.
  * Rituximab will be diluted in an infusion bag of either 0.9% sodium chloride or 5% dextrose.
  * No other drugs will be mixed with it, and patients will be closely monitored for any infusion reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rituximab in treatment refractory Hypersenstivity pneumonitis (Experimental): Patients diagnosed with chronic Hypersensitivity Pneumonitis who have not responded to standard treatment including antigen avoidance and immunosuppressive therapy.
  Interventions: Drug: Rituximab (Mabthera)

INTERVENTIONS:
Drug: Rituximab (Mabthera) — In Chronic hypersensitivity pneumonitis patients with no improvement in lung function (deterioration in their FVC% predicted more than or equal 5%) after a minimum of 6 months treatment including antigen avoidance and immunosuppressive therapy. Rituximab will be administered by an intravenous infusion.
  * Two doses of Rituximab will be given, the first dose at day 0 and the second dose at day 15, 1 gram of Rituximab will be given in each dose.
  * Patients will be given acetaminophen and antihistamine before each infusion.
  * Rituximab will be diluted in an infusion bag of either 0.9% sodium chloride or 5% dextrose.
  * No other drugs will be mixed with it, and patients will be closely monitored for any infusion reactions.

SUMMARY:
Hypersensitivity pneumonitis (HP) presents with a highly variable clinical course, and Traditional treatment involves systemic corticosteroids in conjunction with strict avoidance of the offending antigen. However, a subset of patients with progressive disease remains unresponsive to conventional therapies. The objective of this study is to evaluate the therapeutic potential of Rituximab in individuals with refractory hypersensitivity pneumonitis who did not respond to conventional immunosuppressive therapy and antigen avoidance.

Assessing FVC at three intervals: six months prior to the initiation of Rituximab therapy (M-6), at the time of treatment initiation (M0), and six months afterward (M+6).

DETAILED DESCRIPTION:
The study will be conducted at the Chest Department, Faculty of Medicine, Cairo University during the period between June 2023 to January 2025. This study, which received approval from the Research Ethics Committee of Cairo University code (MD-180-2023), including 30 patients diagnosed with hypersensitivity pneumonitis at the Chest Department, Kasr Al Ainy Hospital, Cairo University.

Inclusion criteria:

1. Age 18 years old and above.
2. Patients with the diagnosis of chronic hypersensitivity pneumonitis, validated during a multidisciplinary team meeting with the criteria adapted from the CHEST guidelines 5, with decline in their FVC of greater than or equal 5% after a minimum of 6 months treatment including antigen avoidance and immunosuppressive therapy (including corticoseroids and Azathioprine).

Exclusion criteria:

1. Hypersensitivity to Rituximab.
2. Severe heart failure.
3. Moderate or severe pulmonary hypertension.
4. Fibrotic hypersensitivity pneumonitis.
5. Pregnancy.
6. Active infection.

Data collection: demographic data of all patients, smoking status, environmental or occupational exposure, onset and duration of symptoms, detailed history of previously received treatment, and oxygen therapy were collected. Assessment of Dyspnea grades using the modified Medical Research Council (mMRC) scale, full clinical examination including assessment of vital signs and chest auscultation were assessed. Routine laboratory investigations (CBC, Coagulation profile, Liver, Kidney functions, ABG) and Serum Immunoglobulins levels before and after initiation of therapy with Rituximab were obtained. All patients were screened for HBV, HCV and HIV infections by measuring hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (anti-HBc), Anti-HCV Antibodies, and Anti-HIV Antibodies. Also, all patients were screened for TB infection using QuantiFERON-TB Gold test. Fiberoptic bronchoscopy with BAL cellular analysis with/without TBLB (transbronchial lung biopsy) together with HRCT were performed to establish the diagnosis of HP and classify the patients into two groups (fibrotic and non-fibrotic). Spirometry and 6 min walk test (6 MWT) were performed to evaluate pulmonary function, Spirometry was performed for each patient three times during the study period, first time was 6 months before immunosuppressive therapy and antigen avoidance (M-6), Second time was at Rituximab administration (M0) and third time was 6 months after Rituximab administration (M+6). Echocardiography was performed to all patients to exclude moderate to severe pulmonary hypertension and heart failure. Prior to Rituximab administration patients were checked for active infection, their vital signs were checked including fever and clinical signs of infection were excluded prior to administration of Rituximab and their laboratory findings including CBC and serum CRP levels were checked to be within normal levels. Two doses of Rituximab were given, the first dose at day 0 and the second dose at day 15, 1 gram of Rituximab was given in each dose by an intravenous infusion. Patients were monitored for symptoms and signs of infections.

Statistical analysis: Data will be collected, tabulated, and statistically analyzed using an IBM compatible personal computer with Statistical Package for the Social Sciences (SPSS) version 26, quantitative data were presented in the form of mean, standard deviation (SD), median and range and qualitative data will be presented in the form numbers (N) and percentages (%), Chi-square test (χ2) or Fisher's Exact test were used to study association between two qualitative variables, Student's t test (t) was used for comparison of quantitative variables between two groups of normally distributed data, Mann-Whitney U test was used for comparison of quantitative variables between two groups of non-normally distributed data, Results will be considered statistically significant at a P value of less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old and above.
2. Patients with the diagnosis of chronic hypersensitivity pneumonitis, validated during a multidisciplinary team meeting with the criteria adapted from the CHEST guidelines, with decline in their FVC of greater than or equal 5% after a minimum of 6 months treatment including antigen avoidance and immunosuppressive therapy (including corticosteroids and Azathioprine).

Exclusion Criteria:

1. Hypersensitivity to Rituximab.
2. Severe heart failure.
3. Moderate or severe pulmonary hypertension.
4. Fibrotic hypersensitivity pneumonitis.
5. Pregnancy.
6. Active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in FVC (% of the predicted value) in chronic hypersensitivity pneumonitis patients 6 months after initiation of Rituximab therapy. | From enrollment to the end of treatment and follow up of the clinical and functional status 18 months
  Forced Vital Capacity (FVC) measured 6 months before rituximab therapy onset (M - 6), at rituximab onset (M0), and 6 months after rituximab intiation (M+6). The FVC% predicted change across treatment time points will be assessed to identify if Rituximab demonstrates potential as an effective treatment for individuals with hypersensitivity pneumonitis unresponsive to conventional therapy.

SECONDARY OUTCOMES:
Change in 6MWD in chronic hypersensitivity pneumonitis patients 6 months after initiation of Rituximab therapy. | From the onset of Rituximab therapy (M0) till 6 months after the onset of therapy (M+6)
  6MWD will be assessed before and after administration of two doses of Rituximab in patients with progressive hypersensitivity pneumonitis who do not respond to antigen avoidance and conventional immunosuppressive therapy
Change in Dyspnea grade by mMRC scale in chronic hypersensitivity pneumonitis patients 6 months after initiation of Rituximab therapy. | From the onset of Rituximab therapy (M0) till 6 months after the onset of therapy (M+6)
  Dyspnea grade by mMRC scale will be assessed before and after administration of two doses of Rituximab in patients with progressive hypersensitivity pneumonitis who do not respond to antigen avoidance and conventional immunosuppressive therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yosri M. Akl, Professor of Chest Diseases, Study Chair — Cairo University; Safy Z. Kaddah, Professor of Chest Diseases, Study Director — Cairo University; Rana K Gabr, MD in Chest Diseases, Principal Investigator — Cairo University; Sherin M. Nassar, MSc in Chest Diseases, Principal Investigator — Cairo University
Locations (1):
- Kasr Al Ainy, Cairo University's Faculty of Medicine, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Akl Y, Kaddah SZ, Nassar SM, El Said RK. Rituximab therapy in patients with treatment-refractory hypersensitivity pneumonitis. Sci Rep. 2025 Oct 17;15(1):36460. doi: 10.1038/s41598-025-21463-y. PMID 41107382